CLINICAL TRIAL: NCT04783935
Title: A 2-year Extension Study to Evaluate Long-term Effectiveness of Mavenclad® in Participants Who Have Completed Trial MS700568_0022 (MAGNIFY MS) (Magnify MS Extension)
Brief Title: Extension to the MAGNIFY MS Trial on Mavenclad® (Magnify MS Extension)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MS700568_0157; 2020-003995-42 (EudraCT Number)
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Mavenclad ®; Cladribine; Relapsing Multiple Sclerosis; Immune cell kinetics
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cladribine

STUDY DESIGN:
Intervention Model Description: Open label, single arm, exploratory, multicenter, 2-year, Phase IV extension study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mavenclad® (Experimental)
  Interventions: Drug: Mavenclad®

INTERVENTIONS:
Drug: Mavenclad® — No intervention was administered as a part of this study. Participants who had received Mavenclad® up to 2 years (Year 1 and 2) in the parent study MS700568_0022 (NCT03364036) were enrolled into this extension study and will be assessed up to 2 years follow-up (Year 3 and 4).
  Other Names: Cladribine

SUMMARY:
The primary purpose of this study was to evaluate the long-term effectiveness of Mavenclad® tablets, in terms of disease activity and safety, in participants with highly-active relapsing multiple sclerosis (RMS) previously participating in the MAGNIFY MS trial MS700568_0022 (NCT03364036).

ELIGIBILITY:
Inclusion Criteria:

* Participants of the MAGNIFY Multiple Sclerosis (MS) trial who received at least a single dose of cladribine tablets during the MAGNIFY MS trial and data on Magnetic resonance imaging (MRI) is available/acquired from at least parent study Month 18 or Month 24 visit and Expanded Disability Status Scale (EDSS) and relapse from parent study Month 24 visit
* Capable of giving signed informed consent

Exclusion Criteria:

* Participant is considered by the Investigator, for any reason, to be an unsuitable candidate for the study
* Participation in other studies/trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (46):
- Australia (2):
  - Liverpool Hospital, Liverpool
  - John Hunter Hospital, New Lambton
- Austria (2):
  - Klinikum Klagenfurt, Klagenfurt
  - Paracelsus Medical University Salzburg, Salzburg
- Canada (4):
  - University of Alberta, Edmonton
  - Children's Hospital, London Health Sciences Centre- Pediatrics, London
  - Montreal Neurological Hospital, Montreal
  - MS Clinical Trials Group, Vancouver
- Czechia (5):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - FN Hradec Kralove, Hradec Králové
  - Nemocnice Pardubickeho kraje, a.s. Pardubicka nemocnice, Pardubice
  - Fakultni nemocnice v Motole, Prague
- Finland (2):
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- France (6):
  - CHU de Montpellier Hôpital Gui de Chauliac- Département de Neurologie, Montpellier
  - CHU Nice - Hôpital Pasteur, Nice
  - CHU Nîmes, Nîmes
  - CHU de Poissy, Poissy
  - CHU de Pontchaillou, Rennes
  - Hôpital Civil, Strasbourg
- Germany (5):
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikum Essen, Essen
  - Neurologische Praxis Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Klinik und Poliklinik fur Neurologie, Leipzig
- Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpo, Szeged, Hungary
- Israel (3):
  - Barzilai Medical Center, Ashkelon
  - Rambam MC, Haifa
  - Sheba Medical Centre, Tel Litwinsky
- Italy (3):
  - Università "G. D'Annunzio" Chieti-Pescara Ospedale Cliniciz, Chieti
  - Dipartimento di internistica clinica e sperimentale "Flaviano Magrassi"Università degli studi della Campania "Luigi Vanvitelli", Napoli
  - IRCSS Neuromed Istituto Neurologico Mediterraneo, Pozzilli
- Poland (3):
  - Samodzielny Publiczny Szpital Kliniczny nr 7 SUM, Katowice
  - Indywidualna Praktyka Lekarska Prof. Konrad Rejdak, Lublin
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 im. Prof. Stanislawa Szyszko SUM w Katowicach, Zabrze
- Spain (5):
  - Hospital de Cruces, Barakaldo
  - Hospital Vithas NISA Sevilla, Castilleja de la Cuesta
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital La Fe, Valencia
- Sweden (2):
  - Sahlgrenska Universitetssjukhus, Gothenburg
  - Akademiskt Specialist Centrum - Centrum för Neurologi,, Stockholm
- United Kingdom (3):
  - Queen Elizabeth Hospital, Birmingham
  - University Hospital of Wales, Cardiff
  - Sheffield Teaching Hospitals Sheffield, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: https://bit.ly/IPD21

REFERENCES:
- [Derived] Schmierer K, Wiendl H, Barkhof F, Montalban X, Achiron A, Derfuss T, Chan A, Hodgkinson S, Prat A, Leocani L, Sellebjerg F, Vermersch P, Jin H, Sponton L, Chudecka A, Gardner L, De Stefano N. Clinical and mechanistic effects of cladribine in relapsing multiple sclerosis: 2-year results from the MAGNIFY-MS Study. Ther Adv Neurol Disord. 2025 Jul 31;18:17562864251351760. doi: 10.1177/17562864251351760. eCollection 2025. PMID 40756532
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS700568_0157
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cladribine: Participants received oral Cladribine (tradename MavencladÂ®) over 2 years, administered as 1 treatment course of 1.75 mg/kg body weight per year in MAGNIFY MS parent study. The treatment course consists of 2 treatment weeks, one at the beginning of the first month and one at the beginning of the second month of the respective treatment year. Each treatment week consists of 4 or 5 days on which a patient receives 10 mg or 20 mg (one or two tablets) as a single daily dose, depending on body weight.
Period: Overall Study
Arm/Group | Cladribine
Started | 219
Completed | 206
Not Completed | 13
Not completed — Withdrawal by Subject | 6
Not completed — PROGRESSIVE DISEASE | 2
Not completed — PATIENT HAS MOVED AND GOES TO ANOTHER HOSPITAL | 1
Not completed — Lost to Follow-up | 3
Not completed — PROTOCOL NON-COMPLIANCE | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cladribine
Number analyzed (Participants) | 219
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142
  Male | 77
Race/Ethnicity, Customized [Number; unit: Participants]
  Ethnicity-Japanese | 0
  Ethnicity-Not Japanese | 204
  Ethnicity-Unknown or Not Reported | 15
  Ethnicity-Hispanic or Latino | 3
  Ethnicity-Not Hispanic or Latino | 201
  Ethnicity-Not Reported | 15
  Race-Asian | 2
  Race-Black or African American | 1
  Race-Other | 6
  Race-Unknown or Not Reported | 26
  Race-White | 184

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With No Evidence of Disease Activity (Three Parameter [NEDA-3]) During Year 3 to 4
Description: The definition of NEDA-3 encompasses a combination of the following 3 related measures of disease activity: No relapses, no confirmed disability progression sustained for 12 weeks as measured on EDSS, and no magnetic resonance imaging (MRI) disease activity, defined as no gadolinium-enhancing (GdE) lesions and no new or enlarging T2 lesions. NEDA-3 was analyzed with the Kaplan-Meier (KM) time-to-event method to reduce the impact of unknown/missing information. EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated. An EDSS progression was defined as an increase of the EDSS score of at least 1.5 point compared to baseline for participants with a baseline EDSS of 0. For participants with an EDSS score between 0.5 and 4.5 at baseline (SD1), EDSS progression was defined as an increase of at least 1 point. For participants with baseline EDSS score of 5, EDSS progression was defined as an increase of at least 0.5.
Time Frame: Year 3 to 4 after the initial dose of Mavenclad® tablets in parent study
Population: The Full Analysis Set included all enrolled, eligible participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cladribine
Number analyzed (Participants) | 219
percentage of participants | 54.23 [47.26 to 60.68]

2. Secondary Outcome: Percentage of Participants With No Evidence of Disease Activity (Three Parameter [NEDA-3]) at Year 3 and at Year 4
Description: as for outcome 1
Time Frame: At Year 3 and 4 after the initial dose of Mavenclad® tablets in parent study
Population: The Full Analysis Set included all enrolled, eligible participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cladribine
Number analyzed (Participants) | 219
percentage of participants
  At Year 3 | 81.63 [75.71 to 86.23]
  At Year 4 | 79.20 [72.30 to 84.56]

3. Secondary Outcome: Percentage of Participants With No Evidence of Disease Activity (Three Parameter [NEDA-3]) After the Start of Study Medication During the Parent Study Until the End of Year 3 and Year 4
Description: as for outcome 1
Time Frame: After the initial dose of Mavenclad® tablets in parent study until the end of Year 3 and 4
Population: The Full Analysis Set included all enrolled, eligible participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cladribine
Number analyzed (Participants) | 219
percentage of participants
  Up to Year 3 | 31.89 [25.81 to 38.11]
  Up to Year 4 | 26.72 [21.03 to 32.74]

4. Secondary Outcome: Percentage of Participants Remaining Three Parameter No Evidence of Disease Activity (NEDA-3) During Year 3 or 4 Among Those With NEDA-3 During Year 1 or 2
Description: as for outcome 1
Time Frame: At Year 3 and 4 after the initial dose of Mavenclad® tablets in parent study
Population: The Full Analysis Set included all enrolled, eligible participants. Number of participants analyzed are number of participants evaluable at that time point in the outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cladribine
Number analyzed (Participants) | 219
percentage of participants
  Year 3 NEDA-3 (During Year 1): number analyzed (Participants) | 72
  Year 3 NEDA-3 (During Year 1) | 92.93 [83.82 to 97.00]
  Year 3 NEDA-3 (During Year 2) | 90.04 [83.47 to 94.09]
  Year 4 NEDA-3 (During Year 1) | 84.86 [72.71 to 91.90]
  Year 4 NEDA-3 (During Year 2): number analyzed (Participants) | 132
  Year 4 NEDA-3 (During Year 2) | 81.92 [72.95 to 88.15]

5. Secondary Outcome: Time to First Disease Activity During Extension Study Period
Description: Time to first disease activity is defined as the time to first occurrence of either qualifying relapse, or 6-month confirmed disability progression (6mCDP), or new or enlarging T2-hyperintense lesions (active T2 lesions), or new T1 Gd+ lesions. The 6MCDP during Extension Study Period is defined as sustained increase in EDSS score that started during the Period. Six-month CDP was considered.
Time Frame: From Month 24 after the initial dose of Mavenclad tablets in parent study until the end of extension study (approximately 2 years)
Population: The Full Analysis Set included all enrolled, eligible participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cladribine
Number analyzed (Participants) | 219
months | 24.05 [19.91 to 24.41]

6. Secondary Outcome: Time to First Disease Activity During up to Parent and Extension Study Period (4 Years)
Description: Time to first disease activity is defined as the time to first occurrence of either qualifying relapse, or 6MCDP, or new or enlarging T2-hyperintense lesions (active T2 lesions), or new T1 Gd+ lesions. The 6MCDP during Extension Study Period is defined as sustained increase in EDSS score that started during the Period. Six-month CDP was considered.
Time Frame: From the initial dose of Mavenclad® tablets in parent study until the end of extension study (approximately 4 years)
Population: The Full Analysis Set included all enrolled, eligible participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cladribine
Number analyzed (Participants) | 219
months | 6.14 [6.05 to 11.70]

7. Secondary Outcome: Time to First New or Enlarging T2 Lesion During Extension Study Period
Description: Time taken for newly enlarging T2 lesions to show up is measured by follow-up MRI.
Time Frame: From the initial dose of Mavenclad® tablets in parent study until the end of extension study (approximately 4 years)
Population: The Full Analysis Set included all enrolled, eligible participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cladribine
Number analyzed (Participants) | 219
months | 6.41 [6.05 to 19.32]

8. Secondary Outcome: Time to First New T1 Gadolinium Enhancing (Gd+) Lesion During Parent and Extension Study Period
Description: Time taken for newly enlarging T1 Gadolinium Enhancing (Gd+) Lesion to show up is measured by follow-up MRI. Kaplan - Meier estimates were used for calculation of data.
Time Frame: From the initial dose of Mavenclad® tablets in parent study until the end of extension study (approximately 4 years)
Population: The Full Analysis Set included all enrolled, eligible participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cladribine
Number analyzed (Participants) | 219
months | NA [50.73 to NA] — Median and upper limit of CI were not calculable due to insufficient number of participants with event across the analysis population during the specified time frame.

9. Secondary Outcome: Time to First Confirmed Disability Progression (CDP) as Measured by Expanded Disability Status Scale (EDSS) During Parent and Extension Study Period
Description: EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated. An EDSS progression was defined as an increase of the EDSS score of at least 1.5 point compared to baseline for participants with a baseline EDSS of 0. For participants with an EDSS score between 0.5 and 4.5 at baseline (SD1), EDSS progression was defined as an increase of at least 1 point. For participants with baseline EDSS score of 5, EDSS progression was defined as an increase of at least 0.5. Kaplan - Meier estimates were used for calculation of data.
Time Frame: From the initial dose of Mavenclad® tablets in parent study until the end of extension study (approximately 4 years)
Population: The Full Analysis Set included all enrolled, eligible participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cladribine
Number analyzed (Participants) | 219
months | NA [NA to NA] — Median and CI were not calculable due to insufficient number of participants with event across the analysis population during the specified time frame.

10. Secondary Outcome: Time to First Qualifying Relapse During Parent and Extension Study Period
Description: A qualifying relapse is defined as new, worsening or recurrent neurological symptoms attributed to Multiple Sclerosis (MS) that last for at least 24 hours without fever or infection, or adverse reaction to prescribed medication, preceded by a stable or improving neurological status of at least 30 days. Kaplan - Meier estimates were used for calculation of data.
Time Frame: From the initial dose of Mavenclad® tablets in parent study until the end of extension study (approximately 4 years)
Population: The Full Analysis Set included all enrolled, eligible participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cladribine
Number analyzed (Participants) | 219
Months | NA [NA to NA] — Median and CI were not calculable due to insufficient number of participants with event across the analysis population during the specified time frame.

11. Secondary Outcome: Time to Recurrent Qualifying Relapse During Parent and Extension Study Period
Description: as for outcome 10
Time Frame: From the initial dose of Mavenclad® tablets in parent study until the end of extension study (approximately 4 years)
Population: The Full Analysis Set included all enrolled, eligible participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cladribine
Number analyzed (Participants) | 219
months | NA [NA to NA] — Median and CI were not calculable due to insufficient number of participants with event across the analysis population during the specified time frame.

12. Secondary Outcome: Time to Treatment Start With Other Disease Modifying Drugs (DMDs) During Parent and Extension Study Period
Description: Time to Treatment Start with Other Disease Modifying Drugs (DMDs) During Parent and Extension Study Period. Kaplan - Meier estimates were used for calculation of data.
Time Frame: From the initial dose of Mavenclad® tablets in parent study until the end of extension study (approximately 4 years)
Population: The Full Analysis Set included all enrolled, eligible participants. As per Protocol, in the parent study, a participant receiving any rescue medication with any other DMD would not participate further in any trial assessments and should have instead completed the early termination visit for final assessment hence no data was collected.
Arm/Group | Cladribine
Number analyzed (Participants) | 0

13. Secondary Outcome: Time to First New or Enlarging T2 Lesion During Extension Study Period
Description: Time taken for newly enlarging T2 Gadolinium Enhancing (Gd+) Lesion to show up is measured by follow-up MRI. Kaplan - Meier estimates were used for calculation of data.
Time Frame: From Month 24 after the initial dose of Mavenclad® tablets in parent study until the end of extension study (approximately 2 years)
Population: The Full Analysis Set included all enrolled, eligible participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cladribine
Number analyzed (Participants) | 219
months | 25.07 [24.41 to NA] — Upper limit of CI were not calculable due to insufficient number of participants with event across the analysis population during the specified time frame.

14. Secondary Outcome: Time to First New T1 Gadolinium Enhancing (Gd+) Lesion During Extension Study Period
Description: as for outcome 8
Time Frame: as for outcome 13
Population: The Full Analysis Set included all enrolled, eligible participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cladribine
Number analyzed (Participants) | 219
months | NA [NA to NA] — Median and CI were not calculable due to insufficient number of participants with event across the analysis population during the specified time frame.

15. Secondary Outcome: Time to First Confirmed Disability Progression (CDP) as Measured by Expanded Disability Status Scale (EDSS) During Extension Study Period
Description: The EDSS is an ordinal clinical rating scale in half-point increments. It assesses the following eight functional systems, areas of the central nervous system that control bodily functions: Pyramidal (ability to walk), Cerebellar (coordination), Brain stem (speech and swallowing), Sensory (touch and pain), Bowel and bladder functions, Visual, Mental, Other (includes any other neurological findings due to Multiple Sclerosis [MS]). EDSS overall score ranging from 0 (normal) to 10 (death due to MS). The 6MCDP during Extension Study Period is defined as sustained increase in EDSS score that started during the Period. Six-month CDP was considered.
Time Frame: as for outcome 13
Population: The Full Analysis Set included all enrolled, eligible participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cladribine
Number analyzed (Participants) | 219
months | NA [NA to NA] — Median and CI were not calculable due to insufficient number of participants with event across the analysis population during the specified time frame.

16. Secondary Outcome: Time to First Qualifying Relapse During Extension Study Period
Description: as for outcome 10
Time Frame: as for outcome 13
Population: The Full Analysis Set included all enrolled, eligible participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cladribine
Number analyzed (Participants) | 219
Months | NA [NA to NA] — Median and CI were not calculable due to insufficient number of participants with event across the analysis population during the specified time frame.

17. Secondary Outcome: Time to Recurrent Qualifying Relapse During Extension Study Period
Description: A qualifying relapse is defined as new, worsening or recurrent neurological symptoms attributed to Multiple Sclerosis (MS) that last for at least 24 hours without fever or infection, or adverse reaction to prescribed medication, preceded by a stable or improving neurological status of at least 30 days.
Time Frame: as for outcome 13
Population: The Full Analysis Set included all enrolled, eligible participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cladribine
Number analyzed (Participants) | 219
months | NA [NA to NA] — Median and CI were not calculable due to insufficient number of participants with event across the analysis population during the specified time frame.

18. Secondary Outcome: Time to Treatment Start With Other Disease Modifying Drugs (DMDs) During Extension Study Period
Description: as for outcome 12
Time Frame: as for outcome 13
Population: as for outcome 12
Arm/Group | Cladribine
Number analyzed (Participants) | 0

19. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a study intervention. A serious adverse event (SAE) was any untoward medical occurrence that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important.
Time Frame: as for outcome 5
Population: The Safety Analysis Set included all participants treated with at least one dose of cladribine tablets during the parent study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cladribine
Number analyzed (Participants) | 219
Participants
  AEs | 142
  Serious AEs | 13

ADVERSE EVENTS:
Time Frame: From Month 24 after the initial dose of Mavenclad tablets in parent study until the end of extension study (approximately 2 years)
Arm/Group | Cladribine
All-Cause Mortality (participants affected / at risk) | 0/219
Serious Adverse Events (participants affected / at risk) | 13/219
Other Adverse Events (participants affected / at risk) | 79/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cladribine (N=219)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Peritonsillitis (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Multiple sclerosis relapse (Nervous system disorders) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cladribine (N=219)
COVID-19 (Infections and infestations) | 50 (50)
Influenza (Infections and infestations) | 11 (11)
Nasopharyngitis (Infections and infestations) | 15 (15)
Upper respiratory tract infection (Infections and infestations) | 12 (12)
Headache (Nervous system disorders) | 16 (16)

LIMITATIONS AND CAVEATS:
The calculation of NEDA-3 rates for single years during the Extension Period (Year 3 and Year 4), may be limited by the sparse measurement of EDSS within each year. This may have resulted in an overestimation of the NEDA-3 rate for each year. In particular, the 6mCDP component requires a confirmatory visit. However, the majority of participants had only 1 visit during each 1-year period, which may have led to an underestimation of the number of events for this component.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT04783935/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT04783935/SAP_001.pdf